CLINICAL TRIAL: NCT03606824
Title: Thyroid Hormone Replacement for Subclinical Hypothyroidism and Dyslipidemia in Patients With Atherosclerotic Cardiovascular Diseases (ThyroHeart-Lipid Study)
Brief Title: Thyroid Hormone Replacement for Subclinical Hypothyroidism and Dyslipidemia in ASCVD (ThyroHeart-Lipid Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaochun.Li (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Peking University Third Hospital (Other); Beijing Chao Yang Hospital (Other); Xuanwu Hospital, Beijing (Other); Beijing Friendship Hospital (Other)
Responsible Party: Sponsor-Investigator, Shaochun.Li, Consultant physician, China National Center for Cardiovascular Diseases
Organization: China National Center for Cardiovascular Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-zx7
Record Dates: First submitted 2018-07-11; First posted 2018-07-31 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Dyslipidemia; Subclinical hypothyroïdism; Statin; ASCVD
Keywords: Thyroid Hormone Replacement; Subclinical Hypothyroidism; Dyslipidemia; ASCVD; Statin
MeSH Terms: conditions — Dyslipidemias | interventions — pitavastatin; Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pivastatin and placebo (Placebo Comparator): After randomization, patients in Pivastatin + placebo group will receive pitavastatin and placebo.
  Interventions: Drug: Pitavastatin and placebo
- Pivastatin and LT-4 (Experimental): After randomization, patients in combination group will receive pitavastatin as the lipid-lowering therapy and take levothyroxine as the thyroid hormone supplement.
  Interventions: Drug: Pitavastatin and levothyroxine

INTERVENTIONS:
Drug: Pitavastatin and placebo — The initial dosage of pitavastatin is 2mg, and it will be regulated according to the level of LDL-C and the upper limit is 4mg.Since the investigators are blind to the arms,the fake regulation of placebo dosage will be same as the Pitavastatin and levothyroxine group.
  Arms: Pivastatin and placebo
Drug: Pitavastatin and levothyroxine — The initial dosage of pitavastatin is 2mg and the initial dosage of levothyroxine is 12.5ug. The dosage of levothyroxine will be regulated according to thyroid function test every 2-3 weeks. The regulation of pitavastatin dosage is same as the monotherapy group.
  Arms: Pivastatin and LT-4

SUMMARY:
In ASCVD patients complicated with subclinical hypothyroidism, the percentage of those who did not reach the target of lipid-lowering therapy (LDL-C>1.8mmol/L) is usually higher than that in population with normal thyroid function. The present study aims to randomly compare two lipid-lowering therapeutic strategies (statins only vs. statins combined with thyroid hormone supplement).

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female;
2. Stable or unstable angina with evidence of myocardial ischemia; coronary angiography reveals stenosis lesions;
3. Subclinical hypothyroidism defined as mild TSH elevation within 5-10mIU/L and normal serum thyroid hormone levels within reference ranges;
4. Level of LDL-C is more than 1.8mmol/L before randomization.
5. Participate in the trial voluntarily and signs the written informed consent form.

Exclusion Criteria:

1. Those who have participated in other drug or therapy equipment clinical trials but did not reach the main study endpoint time limit;
2. Symptoms of severe heart failure (NYHA Class III and above) or left ventricular ejection fraction < 40% (ultrasound or left ventricle ngiography);
3. Pregnant or lactating women;
4. Complicated with severe organ dysfunction: large number of pericardial effusion; acute myocardial infarction; acute myocarditis; acute left heart failure; cardiogenic shock; severe arrhythmia, such as ventricular tachycardia, ventricular fibrillation, frequent atrial / ventricular premature beat, poor control of fast ventricular fibrillation, and bradycardia requiring pacemaker therapy, etc.
5. Patients who are unable to withstand lipid-lowering therapy or thyroid hormone replacement due to allergy to statins or levothyroxine;
6. Serum AST/ALT is three times higher than the upper limits of normal.
7. Patient's life expectancy is less than 12 months;
8. Those waiting for heart transplantation;
9. Patients who are deemed by the researchers to have low compliance and unable to abide by the requirements and complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2019-03-25 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of LDL-C levels | Baseline and 6-month.
  Absolute change value of serum LDL-C levels between the baseline and 6-month assessment.

SECONDARY OUTCOMES:
Changes of non-LDL lipid levels (TC, TG, HDL-C, non-HDL-C) | Baseline and 6-month
  Absolute change value of serum non-LDL lipid levels (including TC, TG, HDL-C, non-HDL-C) between the baseline and 6-month assessment.
LDL-C control rate | Baseline and 1-, 2-, 3- and 6-month assessment.
  Percentages of patients who had LDL-C values below the treatment goal (LDL-C<1.8mmol/L) at 1-, 2-, 3- and 6-month assessment.
Dosage of treatment drugs (pitavastatin and levothyroxine) | At 6-month assessment.
  The dosage of pitavastatin and levothyroxine in combination group at 6-month assessment; The dosage of pitavastatin in control group at 6-month assessment
Levels of thyroid hormones at 6-month assessment | At 6-month assessment.
  Levels of thyroid hormones (thyroid-stimulating hormone, free triiodothyronine, free thyroxine, total triiodothyronine, and total thyroxine) at 6-month assessment
Rates of major adverse cardiac and cerebrovascular events at 6-month assessment | During 6-month follow-up.
  Rates of major adverse cardiac and cerebrovascular events (MACCE, including cardiac death, myocardial infarction, target vessel revascularization and cerebrovascular events) during 6 months follow-up.
Levels of glutamic-pyruvic transaminase (ALT) at 1-, 2-, 3- and 6-month assessment | Baseline and 1-, 2-, 3- and 6-month assessment.
  Safety endpoint: live injury parameters, including levels of glutamic-pyruvic transaminase (ALT) and glutamic-oxaloacetic transaminase (AST).
Levels of glutamic-oxaloacetic transaminase (AST) at 1-, 2-, 3- and 6-month assessment | Baseline and 1-, 2-, 3- and 6-month assessment.
  Safety endpoint: live injury parameters, including levels of glutamic-pyruvic transaminase (ALT) and glutamic-oxaloacetic transaminase (AST).
Levels of serum creatine kinase (CK) at 1-, 2-, 3- and 6-month assessment | Baseline and 1-, 2-, 3- and 6-month assessment.
  Safety endpoint: muscle injury parameter--serum creatine kinase (CK)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Da Tang, MD, Study Chair — Fuwai Hospital, China National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, China National Center for Cardiovascular Diseases, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gjedde S, Gormsen LC, Rungby J, Nielsen S, Jorgensen JO, Pedersen SB, Riis AL, Weeke J, Moller N. Decreased lipid intermediate levels and lipid oxidation rates despite normal lipolysis in patients with hypothyroidism. Thyroid. 2010 Aug;20(8):843-9. doi: 10.1089/thy.2009.0212. PMID 20615126
- [Background] Tzotzas T, Krassas GE, Konstantinidis T, Bougoulia M. Changes in lipoprotein(a) levels in overt and subclinical hypothyroidism before and during treatment. Thyroid. 2000 Sep;10(9):803-8. doi: 10.1089/thy.2000.10.803. PMID 11041458
- [Background] Pazos F, Alvarez JJ, Rubies-Prat J, Varela C, Lasuncion MA. Long-term thyroid replacement therapy and levels of lipoprotein(a) and other lipoproteins. J Clin Endocrinol Metab. 1995 Feb;80(2):562-6. doi: 10.1210/jcem.80.2.7852521.
- [Background] Pearce EN, Wilson PW, Yang Q, Vasan RS, Braverman LE. Thyroid function and lipid subparticle sizes in patients with short-term hypothyroidism and a population-based cohort. J Clin Endocrinol Metab. 2008 Mar;93(3):888-94. doi: 10.1210/jc.2007-1987. Epub 2007 Dec 11. PMID 18073305
- [Background] Lando HM, Burman KD. Two cases of statin-induced myopathy caused by induced hypothyroidism. Endocr Pract. 2008 Sep;14(6):726-31. doi: 10.4158/EP.14.6.726. PMID 18996793
- [Background] Willard DL, Leung AM, Pearce EN. Thyroid function testing in patients with newly diagnosed hyperlipidemia. JAMA Intern Med. 2014 Feb 1;174(2):287-9. doi: 10.1001/jamainternmed.2013.12188. No abstract available. PMID 24217672